CLINICAL TRIAL: NCT01206439
Title: An Advanced Echocardiographic Evaluation of Nebivolol
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Jack Rubinstein (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Jack Rubinstein, Assistant Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC- 09-12-31-04
Record Dates: First submitted 2010-04-02; First posted 2010-09-21 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nebivolol 5 or 10 mg, oral, daily (Experimental): Subject will receive either 5 or 10 mg of oral nebivolol daily. Dose will be determined by control of blood pressure.
  Interventions: Drug: nebivolol

INTERVENTIONS:
Drug: nebivolol — nebivolol 5 or 10 mg oral, daily
  Other Names: Bystolic

SUMMARY:
The purpose of this study is to determine if Nebivolol has any effect on heart function determined by changes in echocardiographic data or exercise tolerance.

DETAILED DESCRIPTION:
Subjects will be given either 5 or 10 mg daily of oral Nebivolol for blood pressure control. They will undergo stress echocardiography at baseline, day 14, 90 and 180.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hypertension
2. Written informed consent before initiation of any study related procedure
3. Baseline Blood pressure > 140 systolic or >90 diastolic if on no antihypertensive therapy.
4. Currently taking one antihypertensive or one antihypertensive and one diuretic for the treatment of hypertension.

Exclusion Criteria:

1. Physical limitations resulting in a limited ability to walk on treadmill for stress echo
2. Intolerance to beta blockers
3. On more than one medication for the treatment of hypertension unless the second medication is a diuretic.
4. Currently pregnant or breast feeding.
5. LFT > 3 X ULN
6. HgA1C > 7
7. Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within past 30 days of enrollment
8. Unwilling to follow protocol or return for study related procedures.
9. Any of the following conditions:

   Coronary artery disease Heart failure Valvular heart disease Ischemic heart disease Atrial fibrillation Pacemaker ICD Hyperlipidemia Diabetes Mellitus Stroke/TIA Anemia COPD Asthma Renal failure requiring dialysis Liver failure Cirrhosis Thyroid dysfunction
10. Any other medical condition that in the PI's opinion could affect myocardial function.
11. Current ETOH or illicit drug abuse -

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Rubinstein, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol 5 or 10 mg, Oral, Daily
Started | 2
Completed | 1
Not Completed | 1
Not completed — subject did not meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nebivolol 5 or 10 mg, Oral, Daily
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic and Diastolic Myocardial Function
Description: Cannot report as only 1 patient was evaluated and data will not be able to remain anonymous.
Time Frame: Baseline to day 180
Population: Insufficient data to analyze.
Arm/Group | Nebivolol 5 or 10 mg, Oral, Daily
Number analyzed (Participants) | 0

2. Secondary Outcome: Exercise Tolerance
Description: Changes in exercise tolerance and time from baseline to 180 days.
Time Frame: Baseline to day 180.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Nebivolol 5 or 10 mg, Oral, Daily
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No